CLINICAL TRIAL: NCT03764774
Title: A Randomized, Placebo-Controlled, Subject- and Investigator-Blind, Single and Multiple Dose, Safety, Tolerability, and Pharmacokinetics Study of LY3463251 in Healthy and Overweight Healthy Subjects
Brief Title: A Study of LY3463251 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial was terminated due to an insufficient benefit/tolerability ratio
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17110; J1D-MC-GZAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- 0.01 Milligram (mg) LY3463251 Part A Cohort 1 (Experimental): Single dose of 0.01 mg LY3463251 administered subcutaneously (SC) on Day 1.
  Interventions: Drug: LY3463251
- 0.03 mg LY3463251 Part A Cohort 2 (Experimental): Single dose of 0.03 mg LY3463251 administered SC on Day 1.
  Interventions: Drug: LY3463251
- 0.1 mg LY3463251 Part A Cohort 3 (Experimental): Single dose of 0.1 mg LY3463251 administered SC on Day 1.
  Interventions: Drug: LY3463251
- 0.3 mg LY3463251 Part A Cohort 4 (Experimental): Single dose of 0.3 mg LY3463251 administered SC on Day 1.
  Interventions: Drug: LY3463251
- 1 mg LY3463251 Part A Cohort 5 (Experimental): Single dose of 1 mg LY3463251 administered SC on Day 1.
  Interventions: Drug: LY3463251
- 3 mg LY3463251 Part A Cohort 6 (Experimental): Single dose of 3 mg LY3463251 administered SC on Day 1.
  Interventions: Drug: LY3463251
- 10 mg LY3463251 Part A Cohort 7 (Experimental): Single dose of 10 mg LY3463251 administered SC on Day 1.
  Interventions: Drug: LY3463251
- 24 mg LY3463251 Part A Cohort 8 (Experimental): Single dose of 24 mg LY3463251 administered SC on Day 1.
  Interventions: Drug: LY3463251
- Placebo Single Dose (Placebo Comparator): Single dose of placebo administered SC.
  Interventions: Drug: Placebo
- 1 mg LY3463251 Part B Cohort 1 (Experimental): 1 mg LY3463251 administered SC, once weekly (QW) for 12 weeks on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
  Interventions: Drug: LY3463251
- 3 mg LY3465231 Part B Cohort 2 (Experimental): 3 mg LY3463251 administered SC, QW for 12 weeks on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
  Interventions: Drug: LY3463251
- 3/6/9 mg LY3463251 Part B Cohort 3 (Experimental): 3 mg LY3463251 administered SC, QW on Days 1 and 8.
  6 mg LY3463251 administered SC, QW on Days 15 and 22.
  9 mg LY3463251 administered SC, QW on Days 29. 36, 43, 50, 57, 64, 71, and 78.
  Interventions: Drug: LY3463251
- 3/9/15/24 mg LY3463251 Part B Cohort (Experimental): 3 mg LY3463251 administered SC, QW on Days 1 and 8.
  9 mg LY3463251 administered SC, QW on Days 15 and 22.
  15 mg LY3463251 administered SC, QW on Days 29 and 36.
  24 mg LY3463251 administered SC, QW on Days 43, 50, 57, 64, 71, and 78.
  Interventions: Drug: LY3463251
- Placebo Multiple Dose (Placebo Comparator): Placebo administered SC, QW for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3463251 — Administered SC
  Arms: 0.01 Milligram (mg) LY3463251 Part A Cohort 1; 0.03 mg LY3463251 Part A Cohort 2; 0.1 mg LY3463251 Part A Cohort 3; 0.3 mg LY3463251 Part A Cohort 4; 1 mg LY3463251 Part A Cohort 5; 1 mg LY3463251 Part B Cohort 1; 10 mg LY3463251 Part A Cohort 7; 24 mg LY3463251 Part A Cohort 8; 3 mg LY3463251 Part A Cohort 6; 3 mg LY3465231 Part B Cohort 2; 3/6/9 mg LY3463251 Part B Cohort 3; 3/9/15/24 mg LY3463251 Part B Cohort
Drug: Placebo — Administered SC
  Arms: Placebo Multiple Dose; Placebo Single Dose

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability (side effects) of single (Part A) and multiple (Part B) doses of the study drug when it is administered subcutaneously (under the skin) into the abdomen.

This is a two-part study. Participants will enroll in only one part. For each participant, Part A will last about 10 weeks and Part B will last about 23 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females

Exclusion Criteria:

* Diagnosed with Type 1 or Type 2 diabetes
* Women who are of childbearing potential or who are breastfeeding
* Donated blood of more than 500 millilitres (mL) within the previous 3 months of study screening
* Have used any tobacco product within 3 months of Day -1, or are unwilling to refrain from the use of tobacco during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benichou O, Coskun T, Gonciarz MD, Garhyan P, Adams AC, Du Y, Dunbar JD, Martin JA, Mather KJ, Pickard RT, Reynolds VL, Robins DA, Zvada SP, Emmerson PJ. Discovery, development, and clinical proof of mechanism of LY3463251, a long-acting GDF15 receptor agonist. Cell Metab. 2023 Feb 7;35(2):274-286.e10. doi: 10.1016/j.cmet.2022.12.011. Epub 2023 Jan 10. PMID 36630958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 4 was terminated early because data from previous cohorts suggested a low probability of achieving competitive weight loss at tolerable doses.
Groups:
- Placebo Single Dose: Single dose of placebo administered subcutaneously (SC) on Day 1
- 0.01 Milligram (mg) LY3463251 Part A Cohort 1: Single dose of 0.01 mg LY3463251 administered SC on Day 1.
- Placebo Multiple Dose: Placebo administered SC, once weekly (QW) on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- 1 mg LY3463251 Part B Cohort 1: 1 mg LY3463251 administered SC, QW on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- 3 mg LY3465231 Part B Cohort 2: 3 mg LY3463251 administered SC, QW on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- 3/6/9 mg LY3463251 Part B Cohort 3: 3 mg LY3463251 administered SC QW on Days 1 and 8.
  6 mg LY3463251 administered SC QW on Days 15 and 22.
  9 mg LY3463251 administered SC QW on Days 29. 36, 43, 50, 57, 64, 71, and 78.
- 3/9/15/24 mg LY3463251 Part B Cohort 4: 3 mg LY3463251 administered SC QW on Days 1 and 8.
  9 mg LY3463251 administered SC QW on Days 15 and 22.
  15 mg LY3463251 administered SC QW on Days 29 and 36.
  24 mg LY3463251 administered SC QW on Days 43, 50, 57, 64, 71, and 78.
Period: Overall Study
Arm/Group | Placebo Single Dose | 0.01 Milligram (mg) LY3463251 Part A Cohort 1 | 0.03 mg LY3463251 Part A Cohort 2 | 0.1 mg LY3463251 Part A Cohort 3 | 0.3 mg LY3463251 Part A Cohort 4 | 1 mg LY3463251 Part A Cohort 5 | 3 mg LY3463251 Part A Cohort 6 | 10 mg LY3463251 Part A Cohort 7 | 24 mg LY3463251 Part A Cohort 8 | Placebo Multiple Dose | 1 mg LY3463251 Part B Cohort 1 | 3 mg LY3465231 Part B Cohort 2 | 3/6/9 mg LY3463251 Part B Cohort 3 | 3/9/15/24 mg LY3463251 Part B Cohort 4
Started | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 13 | 10 | 10 | 18 | 3
Completed | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 6 | 7 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 4 | 11 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 4 | 9 | 0
Not completed — Study Termination | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants, whether or not they completed all protocol requirements.
Groups:
- Placebo Single Dose: Single dose of placebo administered SC on Day 1
- Placebo Multiple Dose: Placebo administered SC, QW on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- 3/9/15/24 mg LY3463251 Part B Cohort 4: 3 mg LY3463251 administered SC, QW on Days 1 and 8.
  9 mg LY3463251 administered SC, QW on Days 15 and 22.
  15 mg LY3463251 administered SC, QW on Days 29 and 36.
  24 mg LY3463251 administered SC, QW on Days 43, 50, 57, 64, 71, and 78.
- Total: Total of all reporting groups
Arm/Group | Placebo Single Dose | 0.01 Milligram (mg) LY3463251 Part A Cohort 1 | 0.03 mg LY3463251 Part A Cohort 2 | 0.1 mg LY3463251 Part A Cohort 3 | 0.3 mg LY3463251 Part A Cohort 4 | 1 mg LY3463251 Part A Cohort 5 | 3 mg LY3463251 Part A Cohort 6 | 10 mg LY3463251 Part A Cohort 7 | 24 mg LY3463251 Part A Cohort 8 | Placebo Multiple Dose | 1 mg LY3463251 Part B Cohort 1 | 3 mg LY3465231 Part B Cohort 2 | 3/6/9 mg LY3463251 Part B Cohort 3 | 3/9/15/24 mg LY3463251 Part B Cohort 4 | Total
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 13 | 10 | 10 | 18 | 3 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (13.9) | 47.0 (18.1) | 52.2 (10.3) | 49.0 (15.8) | 41.0 (17.4) | 35.8 (12.2) | 45.2 (11.5) | 53.8 (2.8) | 43.7 (15.3) | 46.9 (11.6) | 48.2 (11.9) | 45.5 (9.7) | 47.9 (12.4) | 37.0 (10.8) | 46.48 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 3 | 3 | 1 | 0 | 3 | 5 | 1 | 6 | 2 | 4 | 7 | 0 | 43
  Male | 11 | 3 | 3 | 3 | 5 | 6 | 3 | 1 | 5 | 7 | 8 | 6 | 11 | 3 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 5 | 3 | 4 | 5 | 3 | 2 | 3 | 5 | 8 | 8 | 6 | 9 | 3 | 76
  Not Hispanic or Latino | 4 | 1 | 3 | 2 | 1 | 3 | 4 | 3 | 1 | 5 | 2 | 4 | 9 | 0 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 2 | 1 | 4 | 1 | 1 | 0 | 1 | 3 | 2 | 3 | 6 | 2 | 32
  White | 11 | 5 | 4 | 5 | 2 | 4 | 5 | 6 | 5 | 10 | 8 | 7 | 12 | 1 | 85
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 13 | 10 | 10 | 18 | 3 | 118

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Adverse Event(s) (AEs), All Causalities
Description: A summary of serious adverse events (SAEs) and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module
Time Frame: Baseline through follow up in Part A (up to Day 42); Baseline through follow up in Part B (up to Day 123)
Population: All enrolled participants, whether or not they completed all protocol requirements.
Measure: Count of Participants; unit: Participants
Groups:
- 1 mg LY3463251 Part B Cohort 1: 1 mg LY3463251 administered SC, QW for 12 weeks on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- 3 mg LY3465231 Part B Cohort 2: 3 mg LY3463251 administered SC, QW for 12 weeks Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
Arm/Group | Placebo Single Dose | 0.01 Milligram (mg) LY3463251 Part A Cohort 1 | 0.03 mg LY3463251 Part A Cohort 2 | 0.1 mg LY3463251 Part A Cohort 3 | 0.3 mg LY3463251 Part A Cohort 4 | 1 mg LY3463251 Part A Cohort 5 | 3 mg LY3463251 Part A Cohort 6 | 10 mg LY3463251 Part A Cohort 7 | 24 mg LY3463251 Part A Cohort 8 | Placebo Multiple Dose | 1 mg LY3463251 Part B Cohort 1 | 3 mg LY3465231 Part B Cohort 2 | 3/6/9 mg LY3463251 Part B Cohort 3 | 3/9/15/24 mg LY3463251 Part B Cohort 4
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 13 | 10 | 10 | 18 | 3
Participants | 1 | 0 | 0 | 2 | 2 | 2 | 1 | 6 | 6 | 5 | 5 | 5 | 13 | 3

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3463251 Part A
Description: PK: Cmax of LY3463251
Time Frame: Day 1: Predose, 6, 12, 24, 48, 72, 96, 120, 168, 264, 360, 528, 696, and 1008 hr postdose
Population: All participants who received at least one dose of LY3463251 and had evaluable PK data in Part A.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 0.01 Milligram (mg) LY3463251 Part A Cohort 1 | 0.03 mg LY3463251 Part A Cohort 2 | 0.1 mg LY3463251 Part A Cohort 3 | 0.3 mg LY3463251 Part A Cohort 4 | 1 mg LY3463251 Part A Cohort 5 | 3 mg LY3463251 Part A Cohort 6 | 10 mg LY3463251 Part A Cohort 7 | 24 mg LY3463251 Part A Cohort 8
Number analyzed (Participants) | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | NA (NA) — Below quantification level and undetectable, Cmax not calculated. | NA (NA) — Below quantification level and undetectable, Cmax not calculated. | 9.91 (17) | 16.5 (56) | 55.0 (26) | 229 (31) | 583 (35) | 1810 (19)

3. Secondary Outcome: PK: Maximum Observed Concentration of LY3463251 Part B
Description: PK: Cmax of LY3463251
Time Frame: Day 1: Predose, 6, 12, 24, 48, 72, and 120 hours (hr) postdose; Day 8: Predose; Day 15: Predose; Day 28: Predose; Day 57: Predose; Day 78: Predose, and Day 79: 24 hr postdose
Population: All participants who received at least one dose of LY3463251 and had evaluable PK in Part B. Data were not collected for the treatment arms (3 mg and 3/9/15/24 mg) because the study was early terminated prior to participants' assessment at the pre-specified time point (Day 78).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 1 mg LY3463251 QW: 1 mg LY3463251 administered SC, QW on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- 3 mg LY3463251 QW: 3 mg LY3463251 administered SC, QW for 12 weeks on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- 3/6/9 mg LY3463251 QW: 3 mg LY3463251 administered SC, QW on Days 1 and 8.
  6 mg LY3463251 administered SC, QW on Days 15 and 22.
  9 mg LY3463251 administered SC, QW on Days 29, 36, 43, 50, 57, 64, 71, and 78.
- 3/9/15/24 mg LY3463251 QW: 3 mg LY3463251 administered SC, QW on Days 1 and 8.
  9 mg LY3463251 administered SC, QW on Days 15 and 22.
  15 mg LY3463251 administered SC, QW on Days 29 and 36.
  24 mg LY3463251 administered SC, QW on Days 43, 50, 57, 64, 71, and 78.
Arm/Group | 1 mg LY3463251 QW | 3 mg LY3463251 QW | 3/6/9 mg LY3463251 QW | 3/9/15/24 mg LY3463251 QW
Number analyzed (Participants) | 10 | 10 | 18 | 3
ng/mL
  Day 1 | 41.7 (30) | 129 (19) | 150 (38) | 109 (28)
  Day 78: number analyzed (Participants) | 10 | 0 | 18 | 0
  Day 78 | 124 (29) |  | 1190 (15) |

4. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to Time t (AUC [0-tlast]) of LY3463251 Part A
Description: PK: AUC versus time curve from time zero to time t, where t is the last time point with a measurable concentration of LY3463251.
Time Frame: Day 1: Predose, 6, 12, 24, 48, 72, 96, 120, 168, 264, 360, 528, 696, and 1008 hr postdose
Population: All participants who received at least one dose of LY3463251 and had evaluable PK data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram * hour per milliliter (ng*h/mL)
Groups:
- 0.01 mg LY34632515: 0.01 mg LY34632515 on Day 1.
- 0.03 mg LY3463251: 0.03 mg LY3463251 Day 1.
- 0.1 mg LY3463251 Part A: 0.1 mg LY3463251 on Day 1.
- 0.3 mg LY3463251 Part A: 0.3 mg LY3463251 on Day 1.
- 1 mg LY3463251 Part A: 1 mg LY3463251 on Day 1.
- 3 mg LY3463251 Part A: 3 mg LY3463251 on Day 1.
- 10 mg LY3463251 Part A: 10 mg LY3463251 on Day 1.
- 24 mg LY3463251 Part A: 24 mg LY3463251 on Day 1.
Arm/Group | 0.01 mg LY34632515 | 0.03 mg LY3463251 | 0.1 mg LY3463251 Part A | 0.3 mg LY3463251 Part A | 1 mg LY3463251 Part A | 3 mg LY3463251 Part A | 10 mg LY3463251 Part A | 24 mg LY3463251 Part A
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanogram * hour per milliliter (ng*h/mL) | NA (NA) — Below quantification level and undetectable, AUC[0-tlast]) not calculated | NA (NA) — Below quantification level and undetectable, AUC[0-tlast]) not calculated | 1470 (48) | 3010 (50) | 15700 (15) | 75100 (15) | 245000 (17) | 527000 (21)

5. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve During One Dosing Interval (AUC[0-tau)] for LY3463251 Part B
Description: PK: AUC(0-tau) of LY3463251 during one dosing interval on Day 1 and Day 78.
Time Frame: Day 1: Predose, 6, 12, 24, 48, 72, 120, and 168 hours (hr) postdose: Day 78: Predose, 24, 48, 168, 336, 696, 1080 hr postdose
Population: All participants who received at least one dose of LY3463251 and had evaluable PK data in Part B. Data were not collected for the treatment arms (3 mg and 3/9/15/24 mg) because the study was early terminated prior to participants' assessment at the pre-specified time point (Day 78).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- 1 mg LY3465231 Part B: 1 mg LY3465231 SC every week on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- 3 mg LY3465231 Part B: 3 mg LY3463251 administered SC, QW for 12 weeks on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- 3/6/9 mg LY3465231 Part B: 3 mg LY3463251 administered SC, QW on Days 1 and 8. 6 mg LY3463251 administered SC, QW on Days 15 and 22. 9 mg LY3463251 administered SC, QW on Days 29. 36, 43, 50, 57, 64, 71, and 78.
- 3/9/15/24 mg LY3465231 Part B: 3 mg LY3463251 administered SC, QW on Days 1 and 8. 9 mg LY3463251 administered SC, QW on Days 15 and 22. 15 mg LY3463251 administered SC, QW on Days 29 and 36. 24 mg LY3463251 administered SC, QW on Days 43, 50, 57, 64, 71, and 78.
Arm/Group | 1 mg LY3465231 Part B | 3 mg LY3465231 Part B | 3/6/9 mg LY3465231 Part B | 3/9/15/24 mg LY3465231 Part B
Number analyzed (Participants) | 9 | 9 | 18 | 2
ng*h/mL
  Day 1 | 5650 (34) | 18900 (18) | 20400 (41) | NA (NA) — Individual values reported when N = 2: 9810 ng*h/mL, 13700 ng*h/mL
  Day 78: number analyzed (Participants) | 8 | 0 | 7 | 0
  Day 78 | 18000 (33) |  | 167000 (14) |

6. Secondary Outcome: Pharmacodynamics (PD): AUC (0-2hours) of Glucose Part B
Description: AUC of glucose was analyzed using a model with treatment + Day + Treatment*Day + Subject + Random Error where Subject is fitted as a random effect and a repeated statement used with an Unstructured covariance structure.
Time Frame: PD: Day -2; Predose: Day 30 and Day 85 (Part B)
Population: All participants who received at least one dose of LY3463251 and had evaluable PD data in Part B. Data were not collected for the treatment arms (3 mg and 3/9/15/24 mg) because the study was early terminated prior to participants' assessment at the pre-specified time point (Day 85).
Measure: Mean (Standard Deviation); unit: millimole*hour per Liter (mmol*h/L)
Groups:
- Placebo (QW): Placebo administered SC QW on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- 1 mg LY3463251 QW: 1 mg administered SC, QW on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
  .
- 3 mg LY3463251 QW: 3 mg LY3463251 administered SC QW on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- 3/6/9 mg LY3463251 QW: 3 mg LY3463251 administered SC QW on Days 1 and 8.
  6 mg LY3463251 administered SC QW on Days 15 and 22.
  9 mg LY3463251 administered SC QW on Days 29, 36, 43, 50, 57, 64, 71, and 78.
- 3/9/15/24 mg LY3463251 QW: 3 mg LY3463251 administered SC on Days 1 and 8.
  9 mg LY3463251 administered SC on Days 15 and 22.
  15 mg LY3463251 administered SC on Days 29 and 36.
  24 mg LY3463251 administered SC on Days 43, 50, 57, 64, 71, and 78.
Arm/Group | Placebo (QW) | 1 mg LY3463251 QW | 3 mg LY3463251 QW | 3/6/9 mg LY3463251 QW | 3/9/15/24 mg LY3463251 QW
Number analyzed (Participants) | 11 | 9 | 9 | 17 | 3
millimole*hour per Liter (mmol*h/L)
  Day -2 | 14.47 (1.99) | 16.54 (1.95) | 14.04 (3.01) | 15.52 (2.70) | 12.39 (1.72)
  Day 30: number analyzed (Participants) | 10 | 8 | 8 | 8 | 2
  Day 30 | 16.30 (2.39) | 17.37 (2.47) | 17.12 (3.31) | 17.33 (2.78) | NA (NA) — Individual values reported when N=2: 14.73 (3.92) mmol*h/L; 16.38 ( 2.15) mmol*h/L
  Day 85: number analyzed (Participants) | 5 | 8 | 0 | 7 | 0
  Day 85 | 15.64 (2.16) | 15.35 (1.66) |  | 14.51 (2.92) |

7. Secondary Outcome: Change From Baseline in Body Weight at Day 85 Part B
Description: Change from Baseline in Body Weight
Time Frame: Baseline, Day 85 (Part B)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Groups:
- Placebo (QW): Placebo administered SC, QW on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- 3 mg LY3463251 QW: 3 mg LY3463251 administered SC, QW on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
Arm/Group | Placebo (QW) | 1 mg LY3463251 QW | 3 mg LY3463251 QW | 3/6/9 mg LY3463251 QW | 3/9/15/24 mg LY3463251 QW
Number analyzed (Participants) | 13 | 10 | 0 | 18 | 0
kilograms (kg) | 2.11 (1.80) | 0.77 (2.66) |  | -0.28 (2.09) |

ADVERSE EVENTS:
Time Frame: Part A: Baseline up to 42 days Part B: Baseline up to 123 days
Description: All enrolled participants whether or not they completed all protocol requirements.
  Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Placebo: Placebo
- 0.01 mg LY3463251: 0.01 mg LY3463251
- 0.03 mg LY3463251: 0.03 mg LY3463251
- 0.1 mg LY3463251: 0.1 mg LY3463251
- 0.3 mg LY3463251: 0.3 mg LY3463251
- 1 mg LY3463251: 1 mg LY3463251
- 3 mg LY3463251: 3 mg LY3463251
- 10 mg LY3463251: 10 mg LY3463251
- 24 mg LY3463251: 24 mg LY3463251
- Placebo QW: Placebo QW
- 1 mg LY3463251 QW: 1 mg LY3463251 QW
- 3 mg LY3463251 QW: 3 mg LY3463251 QW
- 3/6/9 mg LY3463251 QW: 3/6/9 mg LY3463251 QW
- 3/9/15/24 mg LY3463251 QW: 3/9/15/24 mg LY3463251 QW
Arm/Group | Placebo | 0.01 mg LY3463251 | 0.03 mg LY3463251 | 0.1 mg LY3463251 | 0.3 mg LY3463251 | 1 mg LY3463251 | 3 mg LY3463251 | 10 mg LY3463251 | 24 mg LY3463251 | Placebo QW | 1 mg LY3463251 QW | 3 mg LY3463251 QW | 3/6/9 mg LY3463251 QW | 3/9/15/24 mg LY3463251 QW
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/13 | 0/10 | 0/10 | 0/18 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/13 | 0/10 | 0/10 | 0/18 | 0/3
Other Adverse Events (participants affected / at risk) | 1/16 | 0/6 | 0/6 | 2/6 | 2/6 | 2/6 | 1/6 | 6/6 | 6/6 | 5/13 | 5/10 | 5/10 | 13/18 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=16) | 0.01 mg LY3463251 (N=6) | 0.03 mg LY3463251 (N=6) | 0.1 mg LY3463251 (N=6) | 0.3 mg LY3463251 (N=6) | 1 mg LY3463251 (N=6) | 3 mg LY3463251 (N=6) | 10 mg LY3463251 (N=6) | 24 mg LY3463251 (N=6) | Placebo QW (N=13) | 1 mg LY3463251 QW (N=10) | 3 mg LY3463251 QW (N=10) | 3/6/9 mg LY3463251 QW (N=18) | 3/9/15/24 mg LY3463251 QW (N=3)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 1 (1) | 2 (3) | 10 (14) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hunger (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 6 (10) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (4)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0/5 (0) | 0/3 (0) | 0/3 (0) | 0/3 (0) | 0/1 (0) | 0/0 (0) | 0/3 (0) | 0/5 (0) | 0/1 (0) | 1/6 (1) | 0/2 (0) | 0/2 (0) | 0/7 (0) | 0/0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Cohort 4 was terminated early because data from previous cohorts suggested a low probability of achieving competitive weight loss at tolerable doses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT03764774/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT03764774/SAP_001.pdf